CLINICAL TRIAL: NCT02042066
Title: Efficacy and Safety of Low Intensity- Extracorporeal Shockwave Therapy in Drug Resistant Hypertension
Brief Title: Safety and Efficacy Study of Extracorporeal Shockwave Therapy in the Treatment of Patients With Resistant Hypertension
Acronym: RHT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medispec (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHT-01; 0449-13 (Other: The Department of Clinical Trials - Israel, Hadassah Helsinki Committee)
Record Dates: First submitted 2014-01-19; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Resistant Hypertension; RH; RHT; Blood Pressure; Kidney; Shockwave
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated Group (Experimental): This group will receive actual shockwave treatment
  Interventions: Device: Omnispec model Vascuspec

INTERVENTIONS:
Device: Omnispec model Vascuspec — Energy Density: 0.09 - 0.1 mJ/mm2 Extracorporeal Shockwave Therapy
  Other Names: Vascuspec

SUMMARY:
Low intensity shockwaves have been proven in animal and human studies to increase tissue perfusion, promote angiogenesis and tissue regeneration and improve neural function.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have provided written informed consent.
* Age ≥18 and ≤80 years old.
* Office systolic blood pressure that remains ≥160 mmHg (≥150 mmHg for patient with type 2 diabetes) despite the stable use of ≥3 antihypertensive medications concurrently at maximally tolerated doses, of which one is a diuretic (unless there is a tolerance or a contraindication for a diuretics).
* Able and willing to comply with the required follow-up schedule.

Exclusion Criteria:

* Subjects who have participated in a clinical study involving another investigational drug or device within 4 weeks prior to Screening.
* Have hypertension secondary to an identifiable and treatable cause or take medication that can raise the BP.
* Prior renal artery intervention (balloon angioplasty or stenting).
* Pregnancy.
* Uncompensated heart failure.
* Chronic Liver Disease.
* Patients with skin wound / infection at the treatment area.
* Subjects who take oral anti-coagulants.
* Local tumor of treatment area.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring (ABPM) | 6 Months
  Change in 24 hour ambulatory blood pressure (ABPM) from baseline to six months post last treatment (± 2 weeks)
Ambulatory Blood Pressure Monitoring (ABPM) | 3 Months
  Change in 24 hour ambulatory blood pressure (ABPM) from baseline to three months post last treatment (± 2 weeks)

SECONDARY OUTCOMES:
Office Blood Pressure | 6 Months
  Change in office blood pressure from baseline to three months and six months post last treatment (± 2 weeks).
Serum Urea and Creatinine | 3 Months
  Change in serum urea and creatinine from baseline to 3 months and 6 months (± 2 weeks) post last treatment
Ultrasound | 3 Months
  Change in ultrasound-measured renal resistive index (RRI)
Serum Urea and Creatinine | 6 Months
  Change in serum urea and creatinine from baseline to 3 months and 6 months (± 2 weeks) post last treatment
Adverse Events | 6 Months
Office Blood Pressure | 3 Months
  Change in office blood pressure from baseline to three months and six months post last treatment (± 2 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Shauer, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel